CLINICAL TRIAL: NCT05212779
Title: Predicting the Risk of Ovarian Cancer Recurrence Using Circulating Tumor DNA to Assess Residual Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, John Nakayama, MD, PI, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Other Study IDs: Signatera
Record Dates: First submitted 2021-12-30; First posted 2022-01-28 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual Material for the purpose of validation, quality assurance, and correlation of results, including for regulatory, reimbursement and patent filings, to the extent the foregoing is related or pertains to the results of the research project and the Signatera assay, which is used to perform the research project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Females with Stage II-IV epithelial ovarian cancer: All patients, as participation requirements in this study, are required to have blood drawn at the completion of their adjuvant treatment. Blood sample should be collected within 6 weeks of receiving the last cycle of adjuvant chemotherapy.
  Other optional time points which will be encouraged but not required:
  1. After debulking surgery
  2. Serial draws every 3 months while on maintenance or surveillance.
  Interventions: Diagnostic Test: Signatera testing; Diagnostic Test: Altera Testing

INTERVENTIONS:
Diagnostic Test: Signatera testing — 26mL blood for the first blood draw and tissue sample. 20mL blood all subsequent draws.
Diagnostic Test: Altera Testing — 6ml blood and tissue sample.

SUMMARY:
Blood samples and Tumor tissue will be collected at certain timepoints and will be tested.

DETAILED DESCRIPTION:
Blood samples will be tested by Natera to identify residual tumor DNA for genetic changes in the tumor to potentially improve prediction of long term prognosis and guide treatment options.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of epithelial ovarian cancer stage II-IV

Exclusion Criteria:

Insufficient tumor to perform Signatera testing; Inability to provide consent for the trial

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Epithelial Ovarian Cancer
Study Population: Allegheny Health Network Cancer Institute clinics throughout the system
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of a negative Signatera MRD test on progression free survival (PFS) compared to Signatera MRD testing positive patients. | Signatera MRD testing done within 6 weeks of finishing adjuvant therapy
  The Signatera MRD test measures the amount of circulating tumor DNA(ctDNA). We seek to assess the effect of a negative versus positive test on PFS. PFS will be measured in months from the time of last platinum adjuvant chemotherapy to objective disease progression on imaging according to RECIST 1.1 or death from any cause

SECONDARY OUTCOMES:
To assess the effect of the amount of residual tumor after surgery as defined by Signatera MRD testing on length of PFS | Post debulking surgery
  We seek to assess if the amount of residual tumor detected on Signatera MRD testing correlates with length of PFS. Similarly, does an undetectable ctDNA level versus detectable level (by Signatera MRD testing) have different lengths of PFS. PFS will be measured in months from the time of last platinum adjuvant chemotherapy to objective disease progression on imaging according to RECIST 1.1 or death from any cause.
To assess the effect of negative Signatera MRD testing on the length of overall survival (OS) as compared to Signatera MRD testing positive patients | Signatera MRD testing done within 6 weeks of finishing adjuvant therapy
  This outcomes seeks to assess if a negative Signatera MRD test has a significantly different OS compared to patients with a positive Signatera MRD test. OS will be measured in months from the time of last platinum adjuvant chemotherapy to death from any cause.
To assess the effect of negative Signatera MRD testing on the length of PFS in patients treated with PARP inhibitors (PARPi) compared to Signatera MRD testing positive patients. | Signatera MRD testing done within 6 weeks of finishing adjuvant therapy
  We seek to assess the effect of a negative Signatera MRD test on PFS in patients that are treated with PARPi compared to patients with a positive Signatera MRD test. PFS will be measured in months from the time of last platinum adjuvant chemotherapy to objective disease progression on imaging according to RECIST 1.1 or death from any cause.
To assess if recurrent ovarian cancer is detectable earlier by a rise in ctDNA (by Signatera MRD testing) compared to a rise in CA-125. | Patients will be measured by Signatera MRD testing within 6 weeks of completing adjuvant treatment and every 3 months for up to 2 years. CA-125 will be measured every 3 months until progressive disease or death.
  We seek to assess if Signatera MRD testing will show an increase in ctDNA levels prior to a rise of CA-125 above the normal range.
To assess if recurrent ovarian cancer is detectable earlier by a rise in ctDNA (by Signatera MRD testing) compared to radiographic method (objective disease progression by RECIST 1.1). | Signatera MRD test within 6 weeks of completing adjuvant treatment and every 3 months for up to 2 years. CT every 3 cycles(1 month cycles) while on maintenance or CT for abnormal CA-125, patient symptom, or clinical exam abnormality on surveillance
  We seek to assess if Signatera MRD testing will show an increase in ctDNA levels prior to objective disease progression by RECIST 1.1
To assess if recurrent ovarian cancer is detectable earlier by a rise in ctDNA (by Signatera MRD testing) compared to recurrence as assessed by the investigator. | Patients will be measured by Signatera MRD testing within 6 weeks of completing adjuvant treatment and every 3 months for up to 2 years. Physician assessment wil be as per normal surveillance schedule of the investigator.
  We seek to assess if Signatera MRD testing will show an increase in ctDNA levels prior to the diagnosis of recurrent disease as assessed by physician evaluation. The physician may use all available clinical information in this determination.
To assess the effect of maintenance therapy (PARPi or bevacizumab) on the rate of negative Signatera MRD testing as compared to patients not given maintenance therapy. | Signatera MRD test within 6 weeks of completing adjuvant treatment and every 3 months for up to 2 years.
  We seek to assess if patients will be more likely to achieve a negative Signatera MRD test if they are given maintenance therapy as compared to surveillance.
We seek to determine if patients assessed with whole exome sequencing (Altera) will show different genetic mutational patterns than those who are Signatera MRD testing positive and negative. | Signatera MRD testing done within 6 weeks of finishing adjuvant therapy. Altera testing will be done on the tumor and blood sample provided at enrollment.
  We seek to assess if there are differences in genetic mutations (e.g. BRCA, RAD51, BRIP1, p53, MLH1, PMS2, MSH2 and 6 etc.) between patients that are found to be Signatera MRD testing positive or negative.
We seek to determine if patients assessed with whole exome sequencing (Altera) will show different genetic mutational patterns than those who are PARPi and bevacizumab maintenance therapy responders | Altera testing will be done on the tumor and blood sample provided at enrollment.
  We seek to assess if there are differences in genetic mutations (e.g. BRCA, RAD51, BRIP1, p53, MLH1, PMS2, MSH2 and 6 etc.) between patients that are found to be PARPi and bevacizumab maintenance responders
We seek to determine if patients assessed with whole exome sequencing (Altera) will show different genetic mutational patterns when compared by debulking status. | Altera testing will be done on the tumor and blood sample provided at enrollment.
  We seek to assess if there are differences in genetic mutations (e.g. BRCA, RAD51, BRIP1, p53, MLH1, PMS2, MSH2 and 6 etc.) between patients whose debulking results in no gross residual disease, optimal debulking or suboptimal debulking

CONTACTS AND LOCATIONS:
Overall Officials: John Nakayama, MD, Principal Investigator — Allegheny Health Network
Locations (1):
- AHN West Penn Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No